CLINICAL TRIAL: NCT01814436
Title: Revitalization of Young Immature Permanent Teeth With Necrotic Pulps Using Autologous Stem Cells From Human Exfoliated Deciduous Teeth
Brief Title: Revitalization of Immature Permanent Teeth With Necrotic Pulps Using SHED Cells
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Jin yan, Prof, Professor, Air Force Military Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FourthMMU2013
Record Dates: First submitted 2013-03-16; First posted 2013-03-20 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Dental Pulp Necrosis; Permanent Incisor Avulsed by Trauma
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- scaffold-free SHED-derived pellet (Experimental)
  Interventions: Device: scaffold-free SHED-derived pellet

INTERVENTIONS:
Device: scaffold-free SHED-derived pellet — The purpose of this clinical trial is to both clarify the efficiency of autologous SHED to regenerate pulp and periodontal tissue in the patients with avulsed immature permanent teeth and pulp necrosis to confirm the safety of using autologous stem cells in clinical endodontic regenerative medicine.
  Other Names: SHED pellet

SUMMARY:
Revitalization of Young Immature Permanent Teeth With Necrotic Pulps Using Autologous Stem Cells from Human Exfoliated Deciduous Teeth

DETAILED DESCRIPTION:
Irreversible damage to immature permanent teeth as a result of noxious infection or local trauma before normal physiological closure of the apical structure represents a real clinical challenge. The conventional therapeutic approach is to consider the use of synthetic biocompatible materials, such as calcium hydroxide [Ca(OH)2] and mineral trioxide aggregate (MTA), to induce apical closure, or apexification, by forming a hard tissue barrier across the root apex. However, neither MTA nor calcium hydroxide are currently able either to induce or stimulate pulp regeneration, or to ensure that conventional root development continues once damage has taken place, so that the inherent risk of root fracture remains.

Millions of teeth are accidentally avulsed each year due to the serious trauma in sports, motor vehicle accidents, criminal assaults, and fist fights, among other incidents. The risk is higher in children while their permanent teeth are still immature which may led to lots of complications and also more challenges in treatment. Generally, tooth reimplantation is the most effective therapy for tooth avulsion, As we know, The success of tooth reimplantation depends on the maintenance of vitality of the periodontal ligament, which need the parents and teachers act quickly (e.g., within 2 h) and that the avulsed tooth should preserved in an appropriate medium, such as milk or physiological saline, because the viable cells in the remaining periodontal ligament (PDL) on the root surface play a crucial role in recovering the avulsed tooth functions.

Along with the development of new regenerative protocols to resolve clinical deficiencies, continuing advances in the discovery and characterization of stem cells of dental origin-able to differentiate into multiple tissue types-have recently broadened possible therapeutic horizons towards pulp and periodontal tissue regeneration. Some studies have suggested that the recent discovery and characterization of stem cells from human exfoliated deciduous teeth (SHED) form the cell source of apexogenesis in immature teeth with periradicular periodontitis of endodontic origin. The purpose of this clinical trial is to both clarify the efficiency of autologous SHED to regenerate pulp and periodontal tissue in the patients with immature permanent teeth and pulp necrosis to confirm the safety of using autologous stem cells in clinical endodontic regenerative medicine.

This is a single-centre, randomized, controlled study. This study has been approved by the ethical committees of School of Stomatology, Fourth Military Medical University. The study will be conducted according to the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

1. Those who has signed the informed consent.
2. Those who are between 7-years-old to 12-years-old.
3. Those with at least one young permanent teeth with pulp necrosis which caused by trauma or permanent incisor avulsed by trauma.
4. Those who can provide the health deciduous teeth.
5. Those who have accomplished initial preparation and have been showing good compliance.
6. Those whose guardians understand the purposes of the trial and are capable of making an independent decision to comply with trial requirements
7. Those who are able to visit our hospital in accordance with the trial schedule

Exclusion Criteria:

1. Those in an extremely poor nutritional condition (serum albumin concentration <2 g/dL)
2. Those whose guardians would not cooperate with the treatment.
3. Those who has uncontrollable oral disease.
4. Those with severe dental fear.
5. Those with coexisting mental or consciousness disorder.
6. Those with teeth dysplasia and/or hereditary disease history.
7. Those with systemic disease which may affect the postoperative healing.
8. Those with bruxism and malocclusion.
9. Loss of the avulsed teeth.
10. Those who are taking the medicine which would affect the postoperative healing.
11. Those with the bad oral habits.
12. Those who are undertaking other trail meanwhile or few weeks ago.
13. Those coexisting disease of the blood or immune system.
14. Those who are not capable to provide the deciduous dental pulp cells.
15. Those with the severe tooth trauma (crown-root or root fracture, tooth displacement).
16. Others who the investigators or sub-investigators determined as unsuitable for the trial.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2013-02; Primary Completion 2017-07 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Pulp and Apical regeneration | 1 year following transplantation
  The main outcome measures in the study protocol were: pulp status evaluated by dental pulp vitality tester; pulp revascularization examined by laser dopler flow meter, and the index of clinical examination. In addition, we examined whether and to what extent adverse events, for which causal relationships with the use of SHED cell was not ruled out, emerged.
  The other main outcome measures in the study protocol were: the degree of apical closure; the rate of increase in root length and the change of root canal wall thickness. We examined and evaluate the anatomic morphology of teeth roots using dental computer tomography. We set rate of increase in root length as the most statistically important outcome (primary outcome).

SECONDARY OUTCOMES:
Clinical parameters | 3~12 month following transplantation
  periapical lesion and tooth mobility

CONTACTS AND LOCATIONS:
Overall Officials: songtao shi, PhD, Principal Investigator — chool of Stomatology, Fourth Military Medical Univeristy; Ostrow School of Dentistry, University of Southern California
Locations (1):
- School of Stomatology, Fourth Military Medical University, Xi'an, Shaanxi, China